CLINICAL TRIAL: NCT05239819
Title: The Fully Engaged Inspiratory Muscle Training Reduces Postoperative Pulmonary Complications Rate and Increased Respiratory Muscle Function in Patients With Upper Abdominal Surgery: a Randomized Controlled Trial
Brief Title: The Cardiopulmonary Effects and Diaphragm Function of Complete Inspiratory Muscle Training in Patients With Upper Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Kun-Ling Tsai, Associate Professor, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B-BR-108-012
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Inspiratory Muscle Training; Postoperative Pulmonary Complications; Respiratory Muscle Function; Abdominal Surgery
Keywords: inspiratory muscle training; postoperative pulmonary complications; respiratory muscle function; abdominal surgery
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The study population will be randomized and separated in two groups, Intervention and Usual care group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): We conducted a fully engaged inspiratory muscle training (IMT) program. The exercise group received the intervention threshold IMT from preoperative to postoperative undergoing upper abdominal surgery. The IMT was started before 3 weeks of operation and surveyed in the followed 4 weeks.
  Interventions: Behavioral: Inspiratory muscle training
- Usual care group (Active Comparator): The Usual care group will receive regulated education.
  Interventions: Behavioral: Regulated care and education

INTERVENTIONS:
Behavioral: Inspiratory muscle training — The initial training intensity of the preoperative threshold IMT trainer (DofinTM, Breathing Strength Builder, Taiwan) was moderate to high intensity (≥50% of MIP), which was according to the patient's baseline level and increased by 5-10% per week. The frequency is 25-30 minutes each time, twice a day and five days per week for at least two weeks. The participants would receive at least 10 times training sessions before surgery
  Arms: Intervention group
Behavioral: Regulated care and education — Regulated care and education will be applied
  Arms: Usual care group

SUMMARY:
Upper abdominal surgical treatment may have reduced respiratory muscle function and mucociliary clearance, which might be a consequence of postoperative pulmonary complications (PPCs). The threshold inspiratory muscle training (IMT) may serve as an effective modality to improve respiratory muscle strength and endurance in patients. However, whether this training could help patients with upper abdominal surgery remain to be determined.

ELIGIBILITY:
Inclusion Criteria:

1. ≧20 years old with upper abdominal surgery,
2. American Society of Anesthesiologists; ASA) I-IV
3. body Mass Index; BMI≥ 18
4. able to follow exercise protocol. T

Exclusion Criteria:

1. history of prior abdominal surgery
2. high risk of exercise contraindications (e.g. severe cardiac or cardiovascular disease), 3) American Society of Anesthesiologists; ASA) V-IV

4) unable to follow exercise protocol 5) severe organ failure

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Pulmonary complications rate | Change from baseline (0 week) to follow up (4 weeks)
  According to the definition of PPCs on European Perioperative Clinical Outcome 2015
Respiratory muscles strength | Change from baseline (0 week) to follow up (4 weeks)
  MIP and MEP are done by measuring the upper airway pressure
Diaphragm mobilit | Change from baseline (0 week) to follow up (4 weeks)
  Diaphragm ultrasonography

SECONDARY OUTCOMES:
Quality of life score | Change from baseline (0 week) to follow up (4 weeks)
  The World Health Organization Quality of Life Briefing

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD sharing plan will be decided after summarized data being published

REFERENCES:
- [Derived] Huang YT, Lin YJ, Hung CH, Cheng HC, Yang HL, Kuo YL, Chu PM, Tsai YF, Tsai KL. The fully engaged inspiratory muscle training reduces postoperative pulmonary complications rate and increased respiratory muscle function in patients with upper abdominal surgery: a randomized controlled trial. Ann Med. 2022 Dec;54(1):2222-2232. doi: 10.1080/07853890.2022.2106511. PMID 35942800